CLINICAL TRIAL: NCT03246334
Title: MONITOR-IC: a Mixed Methods Multicenter Prospective Open Cohort Study Determining and Improving Long-term Outcomes of ICU Survivors
Brief Title: MONITOR-IC: Determining and Improving Long-term Consequences of ICU Care
Acronym: MONITOR-IC
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Radboudumc
Record Dates: First submitted 2017-08-02; First posted 2017-08-11 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-08

CONDITIONS: Post-Intensive Care Syndrome (PICS)
Keywords: Cohort study; Critical Care; Follow-up study; Intensive care units; Long-term outcome; Outcome assessment; Quality of life
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Critically ill patients admitted >12 hours to the ICU

SUMMARY:
Due to advances in critical care medicine, more patients survive their critical illness. However, intensive care unit (ICU) survivors often experience long-term physical, cognitive and mental problems, summarized as post intensive care syndrome (PICS), impacting their health related quality of life (HRQoL).

The aims of this study are to study the: 1) long-term outcomes, 2) predictors for PICS, 3) prediction of long-term HRQoL, 4) ratio between HRQoL of ICU-survivors and healthcare related costs, and 5) effects on the long-term of interventions

DETAILED DESCRIPTION:
Specific research questions:

1. What are the post-intensive care symptoms that patients experience after their ICU admissions and what is their HRQoL?
2. What are important predictors for the various physical, cognitive and mental long- term outcomes and health related quality of live outcome, using traditional statistical techniques and sophisticated AI/ML techniques?
3. What is the ratio between HRQoL and healthcare related costs?
4. What are experiences of patients regarding their problems and quality of life after the ICU?
5. What are the effects of interventions aimed to improve long-term outcomes of ICU patients?

Design:

The MONITOR-IC study is an ongoing multicenter prospective open cohort study in which long-term outcomes of ICU patients are studied for a period of two to five years.

The study is carried out in several ICUs in the Netherlands; including academic hospitals, and non-academic hospitals. ICU patients are recruited from July 2016 onwards and followed for two to five years.

Patient recruitment:

Patients scheduled for ICU admission after elective surgery, will be recruited at the outpatient clinic (anaesthesiology or cardiac surgery) (Figure 1). Patients with a non-scheduled admission will be recruited at the ICU. Patients receive information by ICU researchers/nurses/intensivists regarding the aim, content and relevance of the MONITOR-IC, and will be asked for participation. Informed consent is asked for the questionnaires, data from the patients' individual medical record and data from their health insurance company. In case patients are unable to give consent, their legal representative will be asked.

Methods:

Since this is an ongoing open cohort study with multiple questions, several methods will be used including quantitative, qualitatitative and mixed methods.

All patients, or their relatives in case patients are not able to fill in the questionnaire themselves, will be approached to complete the self-administered online questionnaire or on patients' request a paper based: at ICU admission, and several times post-ICU 3 - 12 and 24 months; patients included between 2016 and 2022, also receive the questionnaire 60 months post-ICU. To get insight into the situation before the ICU admission, the baseline questionnaire is provided when the patients are asked for informed consent. This could be preoperatively for the planned admissions or after admission at the ICU. Then, patients are asked to rate their situation before the ICU admission.

Items in questionnaire:

* Patients' health status and HRQoL = SF-12 and the EQ-5D-5L.
* Patients' level of frailty and vulnerability = Clinical Frailty Score (CFS)
* The level of fatigue = CIS-8, a subscale of the Checklist Individual Strength
* Cognitive impairment = abbreviated 14-item Cognitive Failure Questionnaire (CFQ-14).
* Anxiety and depression = Hospital Anxiety and Depression Scale (HADS)
* Subjective distress, caused by traumatic events = Impact of Event Scale 6-questions (IES-6)
* Care needs and support from professionals and informal caregiver
* Social consequences = question set for changes in family circumstances, socio-economic stability and care requirements.

Medical data Patients' demographics and information regarding their diagnosis and treatment, such as primary conditions, pre-existing co-morbidity, disease severity, (re)admission, length of ICU stay, expected mortality (based on the APACHE III-IV models) and medication, will be extracted from their medical record and the Dutch National Intensive Care Evaluation (NICE) registry.

Health Insurance data Healthcare use and related costs, covered by the Dutch healthcare insurance, will be retrieved from Vektis; a Dutch organization which collects and manage health insurance claimed data of all health insurance companies in the Netherlands.This data is collected based on the Diagnosis Treatment Combination (DTC); a total set of activities carried out by the hospital and medical specialists. Additionally, data is collected regarding nursing days, visits at the outpatient clinic and emergency department, nursing homes, ambulance transport, consultation with general practitioner, paramedical care (including physiotherapist, occupational therapist, dietician and speech therapist), prescribed medication, mental healthcare and revalidation. The Vektis database contains data from all for healthcare insured citizens and covers 99% of the total Dutch population. Using patient's unique insurance number the investigators are able to merge patient's insurance data with the questionnaire data and medical data from the medical record at patient level.

Care delivered by community nurses and informal caregivers is not included in the Vektis database and will be studied via the questionnaire.

Interviews To get insight into the patients' experiences post ICU face to face or in case this is not possible, video supported, semi-structured interviews will be conducted with ICU survivors. Interviews will take place at the participants' preferred location (home or clinic, or via video contact).

Patients will be purposively sampled based on various experienced outcomes, such as the quality of life, daily functioning, anxiety, depression, and their experienced needs for more information or emotional support; depending on the research question. Experienced and trained researchers will conduct the interviews. All interviews will be audio recorded and transcribed verbatim.

Analysis Data are been checked on a regular basis to identify out-of-range answers, inconsistent responses, and missing data. Data from the questionnaires, medical record and healthcare insurance data will be merged at patient level. Descriptive statistics will be used to describe baseline characteristics. Depending on the research question, different statististical techniques, including traditional statistical tests, and artificial intelligence/machine learning or deep learning techniques will be used. Subgroups will be identified; supervised (based on their illness and condition e.g. sepsis, delirium, co morbidities, ARDS, length of ICU stay, duration of mechanical ventilation, dialysis, social demographics as age, gender, education, family setting etc) and unsupervised.

Software Package for the Social Sciences (SPSS) or open source R packages will be used for data analysis and for analyzing the interviews Atlas.ti, will be used.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients age 16 years or older;
* admitted at least 12 hours to a trauma, medical, neurosurgery or cardiac surgery ICU;
* gave written informed consent (or by their legal representative).

Exclusion Criteria:

* Patients with a life expectancy of <48 hours;
* receive palliative care;
* are admitted for a donor procedure;
* cannot read and speak the Dutch language;
* or are not able to fill in the questionnaire and do not have family members/ legal representatives either.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients admitted to one of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2050-08 (Estimated); Study Completion 2050-08 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | 2-5 year post-ICU
  SF-12

SECONDARY OUTCOMES:
Health related quality of life | 2 year post-ICU
  EQ5D-5L
Frailty as part of Physical-Cognitive-Mental impairments | 2 year post-ICU
  CFS (Clinical Frailty Score)
Fatigue as part of Physical-Cognitive-Mental impairments | 2 year post-ICU
  CIS-8 (Checklist Individual Strength)
Cognition as part of Physical-Cognitive-Mental impairments | 2-5 year post-ICU
  CFQ-14
Anxiety and depression as part of Physical-Cognitive-Mental impairments | 2 year post-ICU
  HADS (Hospital Anxiety and Depression Scale)
Post traumatic stress disorder as part of Physical-Cognitive-Mental impairments | 2 year post-ICU
  IES-6 (Impact of Event Scale-6 questions)
Patients' care and support needs and social consequences | 2 year post-ICU
  Questionnaire regarding specific needs and supports and social impact post ICU
Patients' healthcare use and related costs | 2 year post-ICU
  Data of healthcare insurance

CONTACTS AND LOCATIONS:
Overall Officials: Mark van den Boogaard, RN, PhD., Principal Investigator — Radboud university medical center, Prof.dr. of Nursing Science in Acute and Critical Care; Marieke Zegers, PhD, Principal Investigator — Radboud university medical center, Senior Researcher dep of Intensive Care Medicine
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porter LL, Hazeleger L, Bos K, Simons KS, van der Hoeven JG, Yeghaian M, van der Woude MCE, van Santen S, Rettig TCD, de Vries M, van den Boogaard M, Zegers M. Identifying distinct clusters of ICU survivors by integrating demographic, pre-admission quality of life, and clinical data: a large prospective cohort study. Intensive Care Med. 2025 Sep;51(9):1603-1614. doi: 10.1007/s00134-025-08052-3. Epub 2025 Aug 7. PMID 40773138
- [Derived] Tilburgs B, Simons KS, Corsten S, Westerhof B, Rettig TCD, Ewalds E, Zegers M, van den Boogaard M. Associations Between Physical, Cognitive, and Mental Health Domains of Post-Intensive Care Syndrome and Quality of Life: A Longitudinal Multicenter Cohort Study. Crit Care Med. 2025 Jan 1;53(1):e74-e86. doi: 10.1097/CCM.0000000000006461. Epub 2024 Oct 24. PMID 39445920
- [Derived] Porter LL, Simons KS, Corsten S, Westerhof B, Rettig TCD, Ewalds E, Janssen I, Jacobs C, van Santen S, Slooter AJC, van der Woude MCE, van der Hoeven JG, Zegers M, van den Boogaard M. Changes in quality of life 1 year after intensive care: a multicenter prospective cohort of ICU survivors. Crit Care. 2024 Jul 25;28(1):255. doi: 10.1186/s13054-024-05036-5. PMID 39054511
- [Derived] van Sleeuwen D, Zegers M, Ramjith J, Cruijsberg JK, Simons KS, van Bommel D, Burgers-Bonthuis D, Koeter J, Bisschops LLA, Janssen I, Rettig TCD, van der Hoeven JG, van de Laar FA, van den Boogaard M. Prediction of Long-Term Physical, Mental, and Cognitive Problems Following Critical Illness: Development and External Validation of the PROSPECT Prediction Model. Crit Care Med. 2024 Feb 1;52(2):200-209. doi: 10.1097/CCM.0000000000006073. Epub 2023 Dec 15. PMID 38099732
- [Derived] Porter LL, Simons KS, Ramjith J, Corsten S, Westerhof B, Rettig TCD, Ewalds E, Janssen I, van der Hoeven JG, van den Boogaard M, Zegers M. Development and External Validation of a Prediction Model for Quality of Life of ICU Survivors: A Subanalysis of the MONITOR-IC Prospective Cohort Study. Crit Care Med. 2023 May 1;51(5):632-641. doi: 10.1097/CCM.0000000000005800. Epub 2023 Feb 20. PMID 36825895
- [Derived] Geense WW, de Graaf M, Vermeulen H, van der Hoeven J, Zegers M, van den Boogaard M. Reduced quality of life in ICU survivors - the story behind the numbers: A mixed methods study. J Crit Care. 2021 Oct;65:36-41. doi: 10.1016/j.jcrc.2021.05.008. Epub 2021 May 23. PMID 34082253
- [Derived] Geense W, Zegers M, Dieperink P, Vermeulen H, van der Hoeven J, van den Boogaard M. Changes in frailty among ICU survivors and associated factors: Results of a one-year prospective cohort study using the Dutch Clinical Frailty Scale. J Crit Care. 2020 Feb;55:184-193. doi: 10.1016/j.jcrc.2019.10.016. Epub 2019 Nov 5. PMID 31739088
- [Derived] Geense W, Zegers M, Vermeulen H, van den Boogaard M, van der Hoeven J. MONITOR-IC study, a mixed methods prospective multicentre controlled cohort study assessing 5-year outcomes of ICU survivors and related healthcare costs: a study protocol. BMJ Open. 2017 Nov 14;7(11):e018006. doi: 10.1136/bmjopen-2017-018006. PMID 29138206